CLINICAL TRIAL: NCT03409588
Title: Treatment of Exercise-Induced Pulmonary Vascular Dysfunction in Symptomatic Patients After Pulmonary Thromboendarterectomy
Brief Title: Treatment of Exercise-Induced Pulmonary Vascular Dysfunction After Pulmonary Thromboendarterectomy or Balloon Pulmonary Angioplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-2349
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Thromboembolic Disease (CTED); Exercise Intolerance Post PEA Surgery
Keywords: Chronic Thromboembolic Disease; CTED; Treatment Post PEA surgery
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Drug (Experimental): Riociguat (Adempas) 0.5mg to 2.5 mg three time daily - oral medication
  Interventions: Drug: Adempas

INTERVENTIONS:
Drug: Adempas — After obtaining baseline data, patients will be placed on oral riociguat at a dose of 0.5 mg TID which will be up titrated over two months to a maximum dose of 2.5 mg TID or maximum tolerated dose. After 3 months from onset of riociguat initiation, the University of California San Diego (UCSD) shortness of breath score, 6 Minute Walk Test (6MWD), and resting/exercise Right Heart Catheterization (RHC) will be repeated.
  Other Names: Riociguat

SUMMARY:
This is an open label study of Riociguat in patients with continued exercise intolerance at least 6 months following pulmonary endarterectomy (PEA).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent PTE or BPA for Chronic thromboembolic pulmonary hypertension (CTEPH) at least six months prior to screening and report ongoing subjective exercise limitation,
* able to give consent
* able to perform a exercise protocol

Exclusion Criteria:

* Patients with known Residual Pulmonary Hypertension (RPH) by RHC following PTE for CTEPH
* ongoing PAH-specific vasodilator therapy
* known contraindication to riociguat
* a physical limitation to completing an exercise protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Change in mean pulmonary arterial pressure | Baseline and 3 months
  Measurements include mPAP (mean pulmonary arterial pressure) measured by right heart catheterization (RHC)
Change in cardiac output | Baseline and 3 months
  Measurements include CO (cardiac output) mPAP/CO slope measured by right heart catheterization (RHC)
Change in Pulmonary artery compliance | Baseline and 3 months
  Measurements include Pulmonary artery compliance measured by right heart catheterization (RHC)

SECONDARY OUTCOMES:
Change in 6 minute walk test | Baseline and 3 months
  Measurements include change in 6 minute walk test (6 MWT) following 3 months of study drug
Change in New York Heart Association (NYHA) functional class | Baseline and 3 months
  Measurements include Change in New York Heart Association (NYHA) functional class following 3 months of study drug
Change in the University of California San Diego (UCSD) shortness of Breath Score | Baseline and 3 months
  Measurements include: Change in the University of California San Diego (UCSD) shortness of Breath Score following 3 months of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bull, MD, Principal Investigator — University of Colorado, Denver; Peter Sottile, MD, Principal Investigator — University of Colorado, Denver; William Cornwell, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No